CLINICAL TRIAL: NCT03967158
Title: Evaluation of Effectiveness and Safety of XIENCE Sierra in Routine Clinical Practice; A MULTICENTER, PROSPECTIVE OBSERVATIONAL STUDY
Brief Title: Evaluation of Effectiveness and Safety of XIENCE Sierra in Routine Clinical Practice
Acronym: IRIS Sierra
Status: Active, not recruiting | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, Professor, Division of Interventional Cardiology. Cardiovascular Center, Asan Medical Center. University of Ulsan, College of Medicine, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2019-03
Record Dates: First submitted 2019-05-27; First posted 2019-05-30 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease; Coronary Disease
Keywords: Xience Sierra; Drug Eluting Stent; Percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Consecutive percutaneous coronary intervention
  Interventions: Device: Xience Sierra stent

INTERVENTIONS:
Device: Xience Sierra stent — Percutaneous coronary intervention with Xience Sierra stent

SUMMARY:
The objective of this study is to evaluate effectiveness and safety of Xience Sierra stent in the "real world" daily practice as compared with other drug-eluting stents.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 and more
* Patient with Xience Sierra Everolimus eluting coronary stent
* Written consent

Exclusion Criteria:

* Intervention with Xience Sierra Everolimus eluting coronary stent and other drug eluting stent at the same time
* Life-expectancy less than 1 year
* Cardiac shock

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with Xience Sierra coronary stent
Sampling Method: Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite event rate of death, non-fatal myocardial infarction (MI), or Target- Vessel Revascularization (TVR) | 1 year

SECONDARY OUTCOMES:
All cause death | 5 year
Cardiac death | 5 year
Myocardial Infarction | 5 year
Composite event rate of death or myocardial infarction (MI) | 5 year
Composite event rate of cardiac death or myocardial infarction (MI) | 5 year
Target- Vessel Revascularization | 5 year
Target- Lesion Revascularization | 5 year
Stent thrombosis | 5 year
Stroke | 5 year
Procedural Success rate | 5 year
  Procedural success rate is defined as < 30 % final stenosis and the absence of in-hospital event including death, myocardial infarction, repeat revascularization.

CONTACTS AND LOCATIONS:
Locations (10):
- South Korea (10):
  - Dong-A Medical Center, Busan
  - Inje University Busan Paik Hospital, Busan
  - Gangwon National Univ. Hospital, Chuncheon
  - Keimyung University Dongsan Medical Center, Daegu
  - Gangneung Asan Hospital, Gangneung
  - Asan Medical Center, Seoul
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul
  - The Catholic University of Korea, Yeouido St. Mary's Hospital, Seoul
  - St.carollo Hospital, Suncheon
  - Wonju Severance Christian Hospital, Wŏnju

IPD SHARING:
Plan to Share IPD: Undecided